CLINICAL TRIAL: NCT05136690
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-over Evaluation of Evoked Responses as Pharmacodynamic Biomarkers in Healthy Adults and Schizophrenic Patients
Brief Title: Evoked Responses as Pharmacodynamic Biomarkers in Healthy and Schizophrenic Participants (MK-4334-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 4334-007; MK-4334-007 (Other: Merck)
Record Dates: First submitted 2021-11-19; First posted 2021-11-29 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Impairment Associated With Schizophrenia
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel A: Healthy Control Participants (Experimental): In Part 1, HC participants receive nicotine patch + capsule placebo, and patch placebo + capsule placebo, under a cross-over design in Periods 1 and 2. In Part 2 (Period 3), HC participants are randomly assigned to receive either MK-4334 250 mg capsule + patch placebo or capsule placebo + patch placebo.
  Interventions: Drug: Nicotine patch; Drug: MK-4334; Drug: Placebo patch; Drug: Placebo capsule
- Panel B: Participants with Mild-to-Moderate SZ (Experimental): In Part 1, participants with mild-to-moderate SZ receive nicotine patch + capsule placebo, and patch placebo + capsule placebo, under a cross-over design in Periods 1 and 2. In Part 2 (Period 3), SZ participants are randomly assigned to receive either MK-4334 250 mg capsule + patch placebo or capsule placebo + patch placebo.
  Interventions: Drug: Nicotine patch; Drug: MK-4334; Drug: Placebo patch; Drug: Placebo capsule

INTERVENTIONS:
Drug: Nicotine patch — Nicotine 21 mg transdermal nicotine patch.
Drug: MK-4334 — MK-4334 250 mg capsule taken by mouth.
Drug: Placebo patch — Placebo patch.
Drug: Placebo capsule — Placebo capsule taken by mouth.

SUMMARY:
The primary purpose of this randomized, double-blind, placebo-controlled cross-over study was to record and measure 40 Hz-auditory steady-state response (ASSR) in healthy controls (HC) and participants with mild-to-moderate schizophrenia (SZ) to determine if the mean inter-trial coherence (ITC) magnitude derived from the 40 Hz-ASSR is lower in SZ than in HC at baseline.

DETAILED DESCRIPTION:
This is a 2-part study. Part 1 was a 2-period study in which participants received either 21 mg nicotine patches and then placebo patches or vice versa, with each patch co-administered with placebo capsules, in a counterbalanced order. In Part 2, participants were randomized to receive either MK-4334 250 mg capsule or placebo capsule, each with placebo patches.

ELIGIBILITY:
Inclusion Criteria:

HC Participants:

* Is in generally good health
* Has no history of clinically relevant neuropsychiatric illness
* Is a mild-to-moderate tobacco user of ≥1-year duration, smoking the equivalent of ~10-15 cigarettes/day

Participants with Mild-to-Moderate SZ:

* Has a current diagnosis of SZ with a duration ≥1 year
* Is clinically stable and in the residual (non-acute) phase of illness for ≥12 weeks prior to the study
* Is stably maintained on a regimen of up to 2 first- or second-generation antipsychotics with no dose changes >50% in combination with concomitant medication commonly prescribed to this population for ≥8 weeks prior to screening and during the study
* Is a mild-to-moderate tobacco user of ≥1-year duration, smoking the equivalent of ~10-15 cigarettes/day

All Participants:

* For males, agrees to be abstinent from heterosexual intercourse, or use an approved contraception method, during the study and for 90 days after the last dose of study drug
* For females, is not of childbearing potential
* Is willing to comply with restrictions on the use of nicotine or nicotine-containing products during the study

Exclusion Criteria:

HC Participants:

* Has known biological family history of psychotic disorder in a first or second degree relative

Participants with Mild-to-Moderate SZ:

* May be excluded from participation by the investigator based on treatment history and/or performance on various screening tests

All Participants:

* Is positive for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV)
* Is at imminent risk of self-harm
* Has had major surgery or donated blood within 4 weeks prior to screening
* Has evidence of cognitive impairment or significant mental disability
* Has a history of clinically significant abnormality or disease
* Has a history of cancer (malignancy)
* Is unable to refrain, or anticipates use, of any non-prescription drugs or herbal remedies
* Has participated in another clinical study within 6 weeks or 5 half-lives (whichever is greater) prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Collaborative Neuroscience Research, LLC ( Site 0002), Long Beach, California
  - Hassman Research Institute Marlton Site ( Site 0001), Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with schizophrenia (SZ) and healthy control (HC) participants were enrolled at 2 study sites in the US.
Groups:
- HC Participants: In Period 1, HC participants received both nicotine patches and placebo patches in a counterbalanced order. All patches were co-administered with placebo capsules. In Period 2, participants received MK-4334 250 mg capsule and placebo capsule in counterbalanced order. All capsules were co-administered with placebo patches.
- Mild-to-Moderate SZ Participants: In Period 1, SZ participants received both nicotine patches and placebo patches in a counterbalanced order. All patches were co-administered with placebo capsules. In Period 2, participants received MK-4334 250 mg capsule and placebo capsule in counterbalanced order. All capsules were co-administered with placebo patches.
Period: Period 1
Arm/Group | HC Participants | Mild-to-Moderate SZ Participants
Started | 13 | 25
Completed | 13 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | HC Participants | Mild-to-Moderate SZ Participants
Started | 13 | 24
Completed | 13 | 20
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Panel A: Healthy Control Participants: In Period 1, HC participants received both nicotine patches and placebo patches in a counterbalanced order. All patches were co-administered with placebo capsules. In Period 2, participants received MK-4334 250 mg capsule and placebo capsule in counterbalanced order. All capsules were co-administered with placebo patches.
- Total: Total of all reporting groups
Arm/Group | Panel A: Healthy Control Participants | Mild-to-Moderate SZ Participants | Total
Number analyzed (Participants) | 13 | 25 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (8.4) | 45.0 (7.8) | 42.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 12 | 22 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 24 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 22 | 32
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Inter-trial Coherence (ITC) Magnitude of 40 Hz-derived Auditory Steady-state Response (ASSR) in HC and SZ Participants at Baseline
Description: The ITC magnitude derived from the 40Hz ASSR is presented. ASSR is measured following a short stream of click trains with a 500 msec inter-train interval (duration), at standard tone and at 40Hz tone. The magnitude of ITC represents the phase consistency of oscillatory activities, in response to EEG coherence at 40Hz stimulation. ITC as a unit of measure is expressed as frequency (40Hz) vs time (msec).
Time Frame: Day -1 (Baseline)
Population: All participants who complied with the protocol sufficiently to ensure the the data are likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Mean (Standard Deviation); unit: ITC (40Hz*msec)
Arm/Group | Panel A: Healthy Control Participants | Mild-to-Moderate SZ Participants
Number analyzed (Participants) | 12 | 25
ITC (40Hz*msec) | 0.432 (0.150) | 0.364 (0.160)

2. Secondary Outcome: Duration Deviant Mismatch Negativity (DD-MMN) in HC and SZ Participants: MMN-A, N100-A, and P3A-A Tests
Description: The mean MMN magnitude derived from baseline DD-MMN will be compared in HC and SZ participants. MMN is measured by subtracting the averaged response to a set of standard stimuli form the average response to deviant stimuli, and taking the amplitude of this difference in a given timepoint. Tests include amplitude of MMN (MMN-A), amplitude of negative peak at 100 msec (N100-A), and amplitude of P3A (P3A-A).
Time Frame: Day -1 (Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Panel A: Healthy Control Participants | Mild-to-Moderate SZ Participants
Number analyzed (Participants) | 13 | 25
µV
  MMN-A Test | -5.207 (2.558) | -3.932 (2.031)
  N100-A Test | -1.616 (1.966) | -1.117 (1.332)
  P3A-A Test | 2.974 (0.774) | 3.121 (1.263)

3. Secondary Outcome: Duration Deviant Mismatch Negativity (DD-MMN) in HC and SZ Participants: MMN-L, N100-L, and P3A-L Tests
Description: The mean MMN magnitude derived from baseline DD-MMN will be compared in HC and SZ participants. The mean MMN magnitude derived from baseline DD-MMN will be compared in HC and SZ participants. MMN is measured by subtracting the averaged response to a set of standard stimuli form the average response to deviant stimuli, and taking the amplitude of this difference in a given timepoint. Tests include latency of MMN (MMN-A), latency of negative peak at 100 msec (N100-A), and latency of P3A (P3A-A).
Time Frame: Day -1 (Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Panel A: Healthy Control Participants | Mild-to-Moderate SZ Participants
Number analyzed (Participants) | 13 | 25
msec
  MMN-A Test | 172.615 (27.122) | 178.880 (25.469)
  N100-A Test | 90.462 (17.704) | 87.680 (14.739)
  P3A-A Test | 284.308 (38.104) | 280.480 (26.691)

4. Secondary Outcome: Effect of Nicotine on Mean ITC Magnitude of 40 Hz-derived ASSR in HC and SZ Participants Compared to Baseline
Description: The effects of nicotine and placebo on in the change from baseline in 40-Hz-derived ASSR were determined in HC and SZ participants on Day 1 or Day 8 in a counterbalanced order, and compared to baseline ASSR. ASSR is measured following a short stream of click trains with a 500 msec inter-train interval (duration), at standard tone and at 40Hz tone. The magnitude of ITC represents the phase consistency of oscillatory activities, in response to EEG coherence at 40Hz stimulation. ITC as a unit of measure is expressed as frequency (40Hz) vs time (msec).
Time Frame: Day -1 (baseline), Day 1, and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ITC (40Hz*msec)
Arm/Group | Panel A: Healthy Control Participants | Mild-to-Moderate SZ Participants
Number analyzed (Participants) | 11 | 23
ITC (40Hz*msec)
  ITC1500 Nicotine: number analyzed (Participants) | 10 | 23
  ITC1500 Nicotine | 0.054 (0.109) | 0.040 (0.043)
  ITC1500 Placebo | 0.000 (0.103) | 0.010 (0.093)

5. Secondary Outcome: Plasma Nicotine Concentration 2 Hours After Patch Application (C2h) Assessed During Event Related Potential (ERP) Recording Sessions
Description: Plasma nicotine levels were determined 2 hours after patch application (C2h) during 21 mg nicotine patch test sessions. Participants received either a nicotine or placebo patch on Days 1 and 8 in a counterbalanced order.
Time Frame: 2 hours after patch application on Day 1 or Day 8
Population: All participants who complied with the protocol sufficiently to ensure the the data are likely to exhibit the effects of treatment, according to the underlying scientific model. Participants received nicotine on either Day 1 or Day 8; results are shown according to actual day of nicotine patch application.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: Healthy Control Participants | Mild-to-Moderate SZ Participants
Number analyzed (Participants) | 2 | 17
nM
  Nicotine on Day 1 | 160.5 (24) | 163.3 (26)
  Nicotine on Day 8: number analyzed (Participants) | 2 | 16
  Nicotine on Day 8 | 119.6 (52) | 159.3 (24)

ADVERSE EVENTS:
Time Frame: Up to approximately 45 days
Description: All treated participants are included. Events are reported according to actual treatment received.
Groups:
- Nicotine 21 mg: All participants who received nicotine 21 mg are included.
- MK-4334 250 mg: All participants who received MK-4334 250 mg are included.
- Placebo: All participants who received placebo are included.
Arm/Group | Nicotine 21 mg | MK-4334 250 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/27 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/27 | 0/38
Other Adverse Events (participants affected / at risk) | 8/37 | 0/27 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine 21 mg (N=37) | MK-4334 250 mg (N=27) | Placebo (N=38)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Application site pruritus (General disorders) | 3 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT05136690/Prot_SAP_000.pdf